CLINICAL TRIAL: NCT05306756
Title: Fetal Scalp Stimulation (FSS) Versus Fetal Blood Sampling (FBS) to Assess Fetal Wellbeing in Labour - a Multi-centre Randomised Controlled Trial.
Brief Title: Fetal Scalp Stimulation Versus Fetal Blood Sampling in Labour
Acronym: FIRSST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient randomizations due to changes in clinical practice
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: University College Cork (Other); University of Limerick (Other); Royal College of Surgeons, Ireland (Other); National University of Ireland, Galway, Ireland (Other); Health Research Board, Ireland (Other); Health Research Board - Trials Methodology Research Network (Other)
Responsible Party: Principal Investigator, Deirdre J Murphy, Professor of Obstetrics, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: DIFA019
Record Dates: First submitted 2022-03-14; First posted 2022-04-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Intrapartum Fetal Distress
Keywords: randomised controlled trial; fetal blood sampling; fetal scalp stimulation; cardiotocography; caesarean section

STUDY DESIGN:
Intervention Model Description: Patients in labor with CTG abnormalities that warrant second-line testing of fetal wellbeing - randomized to digital fetal scalp stimulation (dFSS) versus fetal blood sampling (FBS)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary and perinatal secondary outcomes will be recorded from the computerised delivery record without knowledge of the allocation.
  The principal investigator will play no role in the care of the patient or assessment of outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fetal Blood Sampling (FBS) (Active Comparator): Fetal capillary blood samples will be collected in heparinised tubes and analysed in the delivery suite using the locally available gas analyser. The result of the first technically reliable sample, or the lowest reliable sample if multiple samples are tested, will be interpreted and acted upon according to the protocol, taking account of the clinical circumstances and the stage of labour:
  pH ≥7.25 normal, continue and if indicated repeat in 60 minutes; pH 7.21-7.24 borderline, repeat in 30 minutes; pH ≤ 7.20 abnormal, deliver.
  Interventions: Diagnostic Test: Fetal Blood Sampling (FBS)
- digital Fetal Scalp Stimulation (dFSS) (Active Comparator): The examiner will stimulate the fetal scalp digitally with the index and middle finger over a period of 30-60 seconds.The CTG will be observed over a 5-10 minutes interval after the dFSS and if a fetal heart rate acceleration (>15 bpm for 15 seconds) is observed the test will be considered normal. If there is an episode of normal variability (5-25 bpm) but there is no clear acceleration, the test will be considered borderline. If there is no FHR acceleration and no episode of normal variability with ongoing abnormal features, the test should be interpreted as abnormal in the same way as an abnormal FBS result.
  FHR acceleration normal, if indicated repeat in 60 min; Uncertain acceleration/ normal variability borderline, repeat in 30 minutes; No Acceleration/ongoing abnormal features abnormal, deliver.
  Interventions: Diagnostic Test: digital Fetal Scalp Stimulation (dFSS)

INTERVENTIONS:
Diagnostic Test: Fetal Blood Sampling (FBS) — Vaginal examination, insert amnioscope through cervix, visualise fetal scalp, clean fetal scalp, apply ethyl chloride spray, wipe scalp with petroleum gel, small scalp scratch with sharp instrument, collect sample in heparinised capillary tube, analyse sample.
  Arms: Fetal Blood Sampling (FBS)
Diagnostic Test: digital Fetal Scalp Stimulation (dFSS) — Vaginal examination, insert one or two fingers through cervix onto fetal scalp, rub fetal scalp digitally for approximately 30-60 seconds, withdraw fingers and observe CTG for 5-10 minutes.
  Arms: digital Fetal Scalp Stimulation (dFSS)

SUMMARY:
Pregnant women have routine monitoring of the baby's heart rate when in labour. Women with complicated pregnancies require continuous monitoring using an electronic recorder called a CTG. The CTG produces a paper based recording which is interpreted by the midwife as showing normal, suspicious or abnormal features of the baby's heart rate. Babies quite commonly demonstrate abnormal features from time to time during the course of labour. In some cases the abnormal features are of sufficient concern to warrant delivery by emergency caesarean section. In most of these cases the baby is born in good condition and the question arises whether the caesarean section was unnecessary. In order to reduce the chance of an unnecessary caesarean section additional "second-line" tests can be offered. One such test is where a small drop of blood is taken from the baby's scalp. This test involves an internal examination with an instrument to visualise the baby's head and a small scratch to the baby's scalp. The blood is tested for acid which is an indicator of whether or not the baby is receiving enough oxygen. The test is called a fetal blood sample or FBS. An alternative test is where the doctor or midwife performs a vaginal examination with two fingers and gently rubs the baby's scalp in an attempt to cause an increase in the baby's heart rate. This is a healthy response suggesting that the baby is receiving enough oxygen. The test is called digital fetal scalp stimulation or dFSS. These two "second-line" tests have never been compared in a properly conducted head-to-head comparison. This study aims to compare dFSS and FBS in a large clinical trial completed within four of Ireland's largest maternity hospitals. This trial will generate important evidence of direct relevance to clinical care and patient outcomes.

DETAILED DESCRIPTION:
Continuous electronic fetal heart rate recording with cardiotocography (CTG) is a standard approach to monitoring fetal wellbeing in labour and is recommended for high-risk pregnancies. The aim is to identify fetal compromise early and intervene in order to reduce serious adverse events such as cerebral palsy and perinatal death. CTG abnormalities are relatively common and can lead to the decision to deliver by emergency caesarean section. In most cases the fetus is subsequently found to have been compensating for the stress of labour and is not actually compromised. Fetal blood sampling (FBS) is a second-line invasive test that provides information on the acid-base status of the fetus, reflecting hypoxia. It is used to provide either reassurance that labour can continue, or more objective evidence that delivery needs to be expedited. Clinical guidelines in the United Kingdom and Ireland have treated FBS as a gold standard test. Recent studies have questioned the validity and reliability of FBS, and also the logistic challenges of achieving a result in a timely manner. Fetal scalp stimulation (dFSS) by digital rubbing is an alternative less invasive test of fetal wellbeing in labour and is recommended in preference to FBS in US guidelines. This research aims to compare digital FSS and FBS in women with term singleton pregnancies and an abnormal intrapartum CTG, where additional information on fetal wellbeing is required. A multi-centre randomised controlled trial will be conducted. The clinical outcomes of interest will include caesarean section, assisted vaginal birth, low Apgar scores, cord blood acidosis, and admission to the neonatal unit. This trial will generate important evidence of direct relevance to clinical care and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Singleton pregnancy
* Cephalic presentation
* Gestational age 37+0 weeks or greater
* Abnormal CTG that requires second-line testing (FBS or dFSS)

Exclusion Criteria:

* Contraindication to FBS
* Limited understanding of English
* At the discretion of the responsible obstetrician in cases where there is urgency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Caesarean section (CS) | at birth
  All caesarean sections will be in labour in the context of an abnormal CTG

SECONDARY OUTCOMES:
Caesarean section , primary indication fetal concerns | at birth
  abnormal CTG, or meconium, or low pH on FBS
Caesarean section, primary indication poor progress | at birth
  Poor progress in first or second stage of labour
Caesarean section, failed attempt at assisted vaginal birth | at birth
  Failed vacuum or forceps in second stage of labour
Assisted vaginal birth (AVB) (all cases) | at birth
  Vacuum or forceps or sequential (vacuum and forceps)
Assisted vaginal birth, primary indication fetal concerns | at birth
  abnormal CTG, or meconium, or low pH on FBS
Assisted vaginal birth, primary indication poor progress | at birth
  Poor progress in second stage of labour
Spontaneous Vaginal Birth (SVB) | at birth
  unassisted birth
Decision Delivery Interval (DDI) for emergency CS >30 minutes | during labour up until time of birth
  Decision delivery interval prolonged
Decision Delivery Interval (DDI) for AVB >15 minutes | during labour up until time of birth
  Decision delivery interval prolonged
Perinatal death | up to 7 days of age
  intrapartum or early neonatal death
Late perinatal death | 8-28 days of life
  after 7 days up to 28 days of age
Apgar score at 5 minutes <7 | age 5 minutes
  low Apgar score at 5 minutes
pH umbilical artery <7.00 or Base Excess artery <-12.0 | immediately after birth
  arterial cord blood acidosis
Admission to neonatal unit (NNU) | from birth up until 28 days
  admission all causes
Neonatal encephalopathy (as defined by authors) | from birth up until 28 days
  protocol definition
Therapeutic hypothermia | indicated within 6 hours of birth
  treatment for encephalopathy
Abnormal neurological examination prior to discharge | at time of hospital discharge, assessed up to 28 days after birth
  clinical assessment recording abnormal findings - tone, reflexes, gag
FBS related injury/complication to baby (as reported on neonatal examination) | at birth or with first 7 days of life
  traumatic injury or abnormal bleeding
Major obstetric haemorrhage >1000mL | up to 24 hours after birth
  postpartum haemorrhage
Obstetric Anal Sphincter Injury (OASI - all degrees) | at birth
  injury either spontaneous or with episiotomy
Referral to perinatal mental health services | from birth up to six weeks after birth
  psychological symptoms warranting referral
Maternal acceptability of procedure (defined by questionnaire) | from birth up to 7 days after birth
  acceptability
Number of second-line tests (dFSS or FBS) | during labour up until birth
  each event (rather than samples taken)
Number of inconclusive/uninterpretable dFSS procedures | during labour up until birth
  no clear acceleration or variability borderline
Number of failed FBS procedures | during labour up until birth
  no sample or reliable result achieved

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre J Murphy, MD, Principal Investigator — Trinity College, University of Dublin
Locations (1):
- Coombe Women & Infants University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Subject to request to PI

REFERENCES:
- [Background] Hughes O, Murphy DJ. Comparing second-line tests to assess fetal wellbeing in Labor: a feasibility study and pilot randomized controlled trial. J Matern Fetal Neonatal Med. 2022 Jan;35(1):91-99. doi: 10.1080/14767058.2020.1712704. Epub 2020 Jan 12. PMID 31928269
- [Derived] Yambasu S, Boland F, O'Donoghue K, Curran C, Shahabuddin Y, Cotter A, Gaffney G, Devane D, Molloy EJ, Murphy DJ. Digital Foetal Scalp Stimulation Versus Foetal Blood Sampling to Assess Foetal Well-Being in Labour: A Multicentre Randomised Controlled Trial. BJOG. 2025 Apr;132(5):557-564. doi: 10.1111/1471-0528.18068. Epub 2025 Jan 9. PMID 39780658
- [Derived] Murphy DJ, Shahabuddin Y, Yambasu S, O'Donoghue K, Devane D, Cotter A, Gaffney G, Burke LA, Molloy EJ, Boland F. Digital fetal scalp stimulation (dFSS) versus fetal blood sampling (FBS) to assess fetal wellbeing in labour-a multi-centre randomised controlled trial: Fetal Intrapartum Randomised Scalp Stimulation Trial (FIRSST NCT05306756). Trials. 2022 Oct 4;23(1):848. doi: 10.1186/s13063-022-06794-9. PMID 36195894

DOCUMENTS (1):
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT05306756/ICF_000.pdf